CLINICAL TRIAL: NCT00347399
Title: Effects of Intravitreal Injection of Bevacizumab in Combination With Verteporfin Photodynamic Therapy
Brief Title: Bevacizumab and Photodynamic Therapy in Neovascular Age Related Macular Degeneration
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: undefined
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AvastinTFD
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Age Related Macular Degeneration
Keywords: macular degeneration; antibodies; angiogenesis inhibitor
MeSH Terms: conditions — Macular Degeneration | interventions — Bevacizumab

INTERVENTIONS:
Drug: bevacizumab intravitreal injection
Procedure: verteporfin photodynamic therapy

SUMMARY:
The purpose of this study is to determine if of combination therapy of intravitreal bevacizumab 4 days after the application of photodynamic therapy could improve the visual outcomes of patients with neovascular age related macular degeneration.

DETAILED DESCRIPTION:
The neovascular age related macular degeneration(AMD) is a important cause of legal blindness in adults older than 50 years. Currently the treatment is photodynamic therapy that offer stabilization and limited visual improvement after 2 years of therapy. Bevacizumab has been reported effective used as intravenous injection for AMD. But serious side effects have been reported with the use of this drug in oncologic patients. The intravitreal use has been reported in limited case reports and safety and efficacy should be determined. The purpose of this study is efficacy and safety of 2.5 mg intravitreal of bevacizumab for AMD 4 days after photodynamic therapy with verteporfin

ELIGIBILITY:
Inclusion Criteria:

55 years old neovascular Age related acular degeneration subfoveolar neovascular membrane best corrected visual acuity better than 20/200 snellen (1.0 logMAR)

Exclusion Criteria:

* Previously treated eyes glaucoma diabetes mellitus uncontrolled hypertension coronary artery disease

Ages: 55 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-03 (Actual); Primary Completion 2006-06-30 (Actual); Study Completion 2007-06-30 (Actual)

PRIMARY OUTCOMES:
Visual acuity improvement at 6 months | undefined
  undefined

SECONDARY OUTCOMES:
Retinal thickness improvement at 6 months | undefined
  undefined

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Quiroz-Mercado, MD, Study Director — Asociación para Evitar la Ceguera en México; Jose Dalma Weizhaus, MD, Principal Investigator — Asociación para Evitar la Ceguera en México
Locations (1):
- Hospital Luis Sanchez Bulnes, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Rosenfeld PJ, Moshfeghi AA, Puliafito CA. Optical coherence tomography findings after an intravitreal injection of bevacizumab (avastin) for neovascular age-related macular degeneration. Ophthalmic Surg Lasers Imaging. 2005 Jul-Aug;36(4):331-5. PMID 16156152